CLINICAL TRIAL: NCT06778915
Title: Refining Surgical Strategies Based on Tumor Staging in Head and Neck Adenoid Cystic Carcinoma: Evidence from a Retrospective Cohort Study
Brief Title: Surgical Strategy for Head and Neck Adenoid Cystic Cancer
Status: Completed | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Guopei Zhu, Principal Investigator, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Other Study IDs: 2024HNRT02
Record Dates: First submitted 2025-01-09; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Adenoid Cystic Carcinoma
MeSH Terms: conditions — Carcinoma, Adenoid Cystic | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: surgery — surgery

SUMMARY:
To investigate the relationship between surgical margins and outcomes across different tumor stages, in order to provide evidence and guidance for refining stage-specific surgical approaches.

DETAILED DESCRIPTION:
Adenoid cystic carcinoma of the head and neck (HNACC) presents unique surgical challenges due to its propensity for perineural spread and proximity to critical craniofacial structures. While surgical resection remains the cornerstone of treatment, determining the optimal extent of resection to balance oncologic control and functional preservation requires further investigation. The investigator aimed to investigate the relationship between surgical margins and outcomes across different tumor stages, in order to provide evidence and guidance for refining stage-specific surgical approaches.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent surgical resection with curative intent and PORT.

Exclusion Criteria:

* underwent only biopsy, presented with distant metastases or second primary malignancies at initial diagnosis, had incomplete clinical or histopathologic data, or had histologic evidence of high-grade transformation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: head and neck adenoid cystic carcinoma
Sampling Method: Probability Sample
Enrollment: 309 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Local control | 5 year
  defined as the absence of tumor persistence, recurrence, or progression at the primary tumor site following the completion of treatment, assessed by clinical examination and imaging at designated follow-up intervals.

SECONDARY OUTCOMES:
Locoregional Recurrence-Free Survival (LRRFS) | 5 year
  time from treatment initiation to either locoregional recurrence or death from any cause
Overall Survival (OS) | 5 year
  time from treatment initiation to death from any cause
Distant Metastasis-Free Survival (DMFS) | 5 year
  time from treatment initiation to either distant metastasis or death from any cause

IPD SHARING:
Plan to Share IPD: No